CLINICAL TRIAL: NCT03185377
Title: The Study of Early Detection, Disease Course and Prognosis of Pulmonary Thromboembolism in Chronic Pulmonary Hypertension
Brief Title: Registry for Chronic Obstructive Pulmonary Disease With Pulmonary Thromboembolism in China
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Chinese Academy of Medical Sciences, Fuwai Hospital (Other)
Responsible Party: Principal Investigator, Jianguo He, Chief of Pulmonary Vascular Disease Center, Chinese Academy of Medical Sciences, Fuwai Hospital
Other Study IDs: 2016YFC1304402A
Record Dates: First submitted 2017-06-11; First posted 2017-06-14 (Actual); Last update posted 2017-06-14 (Actual); Status verified 2017-06

CONDITIONS: COPD; PTE - Pulmonary Thromboembolism
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Pulmonary Embolism

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Biospecimen Retention: Samples With DNA — Serum and blood cell
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Chronic obstructive pulmonary disease (COPD) is closely related to venous thromboembolism (VTE). But it is difficult to identify VTE in COPD patients in clinical practice. Therefore, the prevalence data of PTE in COPD is limited. Pulmonary thromboembolism (PTE) is an important factor effecting patients outcomes, but existing researches only have short follow-up time less than 1 year. This study aim to develop an early detection system of PTE in COPD and explore the disease course and prognosis.

ELIGIBILITY:
Inclusion Criteria:

* Patients hospitalized for chronic obstructive pulmonary disease (COPD) exacerbation

Exclusion Criteria:

* Stable COPD patients
* COPD hospitalized for definite causes other than pulmonary thromboembolism
* Patients with malignant tumor
* Patients with contraindications for CT pulmonary angiography
* Psychopath

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: COPD patients
Sampling Method: Non-Probability Sample
Enrollment: 1708 (Estimated)
Dates: Start 2017-03-15 (Actual); Primary Completion 2020-12-31 (Estimated); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
All-cause mortality | 3 years
  mortality in %

SECONDARY OUTCOMES:
COPD exacerbations | 3 years
  Total times
venous thromboembolism recurrence | 3 years
  total times
major bleeding | 3 years
  total times

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Chaoyang Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided